CLINICAL TRIAL: NCT05620264
Title: Validation of Interleukins and Other Cytokines Together With OCT Imaging for Rapid Infectious Keratitis Assessment
Acronym: VICTORIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-002
Record Dates: First submitted 2022-10-05; First posted 2022-11-17 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Keratitis Bacterial; Keratitis Fungal
Keywords: Keratitis; Optical Coherence Tomography; Cytokine Quantification; Tear Film
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Tear Film
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Keratitis Group: Patients with clinically suspected bacterial or fungal keratitis
  Interventions: Diagnostic Test: Tear Sample Probe

INTERVENTIONS:
Diagnostic Test: Tear Sample Probe — Samples will be collected by conjunctival lavage of the affected eye without topical anesthesia. Sterile normal saline will be infused at room temperature into the lower conjunctival sac by gently pulling down the lower eyelid and with a needle-free insulin syringe. After few seconds, the lavage fluid will be aspirated back into the same syringe without the syringe touching the conjunctiva.

SUMMARY:
As conventional corneal scraping with bacterial culturing has several disadvantages such as long duration until diagnosis, invasiveness and lacks alternatives, there is demand for a novel non-invasive, rapid test in keratitis management. First aim of this study will be to evaluate the influence of TNF-alpha on Gram+ and Gram- bacteria causing keratitis. Second aim of this study will be to develop an algorithm, that should help to distinguish between different pathogens causing keratitis.

DETAILED DESCRIPTION:
Infectious or inflammatory processes of the cornea (keratitis) are common and vision threatening. They are the 5th leading cause of blindness and especially infectious keratitis is responsible for 2,000,000 new blind eyes per year (worldwide). Commonly, the presence and nature of bacterial pathogens is determined by taking scratches from the cornea, subsequent Gram stain and examination of microbiological cultures. Major problems in therapeutic decision-making pose the long duration of bacterial culturing for pathogen detection (approximately one week), relatively low sensitivity and increasingly frequent bacterial resistances to antibiotic agents.

In small previous studies optical coherence tomography (OCT) combined with analysis of tear cytokines were found to be supportive in distinguishing between different pathogens causing keratitis. These studies appear to be a game changer in the field of rapid testing for keratitis. However, the problem of these studies is a small sample size and the use of partially outdated equipment.

Benefit/risk assessment Although there is no direct benefit for participating subjects, the results of the study can help to gain more insight into the course of keratitis and could further improve the diagnostic utilities in disease management.

There is no additional medication used in this study. The findings of the present study could help to establish a better understanding of keratitis and could enable faster and target-oriented therapy. All applied measurement techniques are painfree.

Thus, the risk to benefit ratio seems to be acceptable.

Study objectives

Primary:

• Comparison of TNF-alpha level differences in tear film (pg/ml) between Gram+ and Gram- bacteria causing keratitis (z test for non-paired samples).

Secondary:

* To develop an algorithm, that should help to distinguish between different pathogens causing keratitis using cytokine levels and OCT findings. This part of the study will be experimental (partial least squares regression and regression random forest plots)
* Levels of IL-1alpha, IL-1beta, IL-6, IL-8, IL-10, IL-17A, TNF-alpha in keratitis
* Morphological findings in optical coherence tomography: corneal thickness (µm), infiltrate thickness (µm), reflectivity of the infiltrate (grey level, where 0 is black and 255 is white).

Design: Prospective single center trial The participants will be recruited from the ambulances of Kepler University clinic, ophthalmology, Linz, Austria A total of 392 patients will be included in this study. Aimed power: 0.8 significance level after a Bonferroni correction for 7 explanatory variables (7 different cytokines): 0.07 Used values (TNF alpha 2): Group 1: 18.8 (26.36) and Group 2: 50.12 (103.83) Parameters Results Power 0.800 alpha 0.007 Mean (Group 1) 18.8 Mean (Group 2) 50.12 Std. deviation (Group 1) 26.36 Std. deviation (Group 2) 103.83 Sample size 1 146 Sample size 2 146 Power (obtained) 0.798 For correction of a potential rounding error (calculated power 0.798) one case should be added to each group.

Although there will not be any study follow-ups the investigator still expects a drop-out rate of 30% for the following reason: As published previously, 67% of all corneal biopsies result in a positive culture. 13 In those cases, where the culture does not provide positive results, the patient will have to be excluded from the analysis.

Therefore, the investigator will include 147 + 147 + (147+147)*0.33 = 391.02 eyes -> 392 eyes Analysis of data is only possible, if the corneal biopsy is positive (a pathogen causing the keratitis is found). Therefore, the investigator expects that approximately 30% of the patients will not be included for analysis. In these cases, the OCT images will still be evaluated, but the tear film sample will be either disposed according to the protocol of tissue waste or if the investigating ophthalmologist expects a non-infectious type of keratitis (such as a neurotrophic ulcer) the cytokine quantification will be performed.

Measurement techniques CASIA 2 (Tomey, Japan) is a ss-OCT biometer that allows high resolution imaging of the anterior segment of the eye.

Tear sampling and cytokine analysis Samples will be collected by conjunctival lavage of the affected eye without topical anesthesia. Sterile normal saline will be infused at room temperature into the lower conjunctival sac by gently pulling down the lower eyelid and with a needle-free insulin syringe. After few seconds, the lavage fluid will be aspirated back into the same syringe without the syringe touching the conjunctiva. Afterwards, the sample will be stored at -80° Celsius until all samples are collected. As mentioned in those samples, where the corneal biopsy was negative, will either be disposed, or (if the ophthalmology expects a non-infectious type of keratitis) still be analysed. Therefore, the conjunctival fluid from the syringes will be pooled and spun down in a centrifuge (400xg for 10 min at 4°C). The Supernatants will be analyzed using the pro-inflammatory multiplex assay kit from Meso Scale Discovery (Gaithersburg, MD, USA) for levels of the following cytokines and chemokines: IL-1alpha, IL-1beta, IL-6, IL-8, IL-10, IL-17A, TNF-alpha. Eighty samples will be analysed at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age of at least 18 years to 119 years
* Written informed consent prior to study-related procedures
* First presentation with keratitis (corneal epithelial ulceration, corneal edema and/or stromal infiltration with inflammatory cells) within 10 days.
* Untreated keratitis or keratitis not responding to the given treatment

Exclusion Criteria:

Subjects will be excluded if one or more of the following criteria apply:

* Symptoms for more than 10 days
* Presence or history of a severe medical condition as judged by the clinical investigator
* Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 119 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the ambulances of Kepler University clinic, ophthalmology, Linz, Austria
Sampling Method: Non-Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
TNF Alpha in Tear Film | The measurement is assessed at the point of study inclusion.
  Comparison of TNF-alpha level differences in tear film between Gram+ and Gram- bacteria causing keratitis

SECONDARY OUTCOMES:
Interleukins | The measurement is assessed at the point of study inclusion.
  Levels of IL-1alpha, IL-1beta, IL-6, IL-8, IL-10, IL-17A
Anterior segment Optical Coherence Tomography | The measurement is assessed at the point of study inclusion
  Morphological findings in optical coherence tomography: corneal thickness, infiltrate thickness, reflectivity of the infiltrate

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — JKU Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
If IPD is going to be shared, is still in evaluation and will be decided throughout the study.

REFERENCES:
- [Background] Ting DSJ, Ho CS, Deshmukh R, Said DG, Dua HS. Infectious keratitis: an update on epidemiology, causative microorganisms, risk factors, and antimicrobial resistance. Eye (Lond). 2021 Apr;35(4):1084-1101. doi: 10.1038/s41433-020-01339-3. Epub 2021 Jan 7. PMID 33414529
- [Background] Konstantopoulos A, Cendra MDM, Tsatsos M, Elabiary M, Christodoulides M, Hossain P. Morphological and cytokine profiles as key parameters to distinguish between Gram-negative and Gram-positive bacterial keratitis. Sci Rep. 2020 Nov 18;10(1):20092. doi: 10.1038/s41598-020-77088-w. PMID 33208864
- [Background] Konstantopoulos A, Del Mar Cendra M, Tsatsos M, Elabiary M, Christodoulides M, Hossain P. Author Correction: Morphological and cytokine profiles as key parameters to distinguish between Gram-negative and Gram-positive bacterial keratitis. Sci Rep. 2021 Feb 26;11(1):5168. doi: 10.1038/s41598-021-85007-w. No abstract available. PMID 33637814
- [Background] Chodosh J, Astley RA, Butler MG, Kennedy RC. Adenovirus keratitis: a role for interleukin-8. Invest Ophthalmol Vis Sci. 2000 Mar;41(3):783-9. PMID 10711694
- [Background] Peng L, Zhong J, Xiao Y, Wang B, Li S, Deng Y, He D, Yuan J. Therapeutic effects of an anti-IL-6 antibody in fungal keratitis: Macrophage inhibition and T cell subset regulation. Int Immunopharmacol. 2020 Aug;85:106649. doi: 10.1016/j.intimp.2020.106649. Epub 2020 Jun 5. PMID 32504999
- [Background] Vasanthi M, Prajna NV, Lalitha P, Mahadevan K, Muthukkaruppan V. A pilot study on the infiltrating cells and cytokine levels in the tear of fungal keratitis patients. Indian J Ophthalmol. 2007 Jan-Feb;55(1):27-31. doi: 10.4103/0301-4738.29491. PMID 17189883
- [Background] Zhang Y, Liang Q, Liu Y, Pan Z, Baudouin C, Labbe A, Lu Q. Expression of cytokines in aqueous humor from fungal keratitis patients. BMC Ophthalmol. 2018 Apr 19;18(1):105. doi: 10.1186/s12886-018-0754-x. PMID 29673332
- [Background] Azher TN, Yin XT, Stuart PM. Understanding the Role of Chemokines and Cytokines in Experimental Models of Herpes Simplex Keratitis. J Immunol Res. 2017;2017:7261980. doi: 10.1155/2017/7261980. Epub 2017 Apr 9. PMID 28491875
- [Background] Wang L, Wang R, Xu C, Zhou H. Pathogenesis of Herpes Stromal Keratitis: Immune Inflammatory Response Mediated by Inflammatory Regulators. Front Immunol. 2020 May 13;11:766. doi: 10.3389/fimmu.2020.00766. eCollection 2020. PMID 32477330
- [Background] Song XJ, Li DQ, Farley W, Luo LH, Heuckeroth RO, Milbrandt J, Pflugfelder SC. Neurturin-deficient mice develop dry eye and keratoconjunctivitis sicca. Invest Ophthalmol Vis Sci. 2003 Oct;44(10):4223-9. doi: 10.1167/iovs.02-1319. PMID 14507865
- [Background] Cole N, Bao S, Willcox M, Husband AJ. Expression of interleukin-6 in the cornea in response to infection with different strains of Pseudomonas aeruginosa. Infect Immun. 1999 May;67(5):2497-502. doi: 10.1128/IAI.67.5.2497-2502.1999. PMID 10225913
- [Background] Cole N, Krockenberger M, Stapleton F, Khan S, Hume E, Husband AJ, Willcox M. Experimental Pseudomonas aeruginosa keratitis in interleukin-10 gene knockout mice. Infect Immun. 2003 Mar;71(3):1328-36. doi: 10.1128/IAI.71.3.1328-1336.2003. PMID 12595449
- [Background] Diamond J, Leeming J, Coombs G, Pearman J, Sharma A, Illingworth C, Crawford G, Easty D. Corneal biopsy with tissue micro-homogenisation for isolation of organisms in bacterial keratitis. Eye (Lond). 1999 Aug;13 ( Pt 4):545-9. doi: 10.1038/eye.1999.135. PMID 10692928